CLINICAL TRIAL: NCT05332067
Title: Omalizumab Before Onset of Exacerbations
Acronym: OBOE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, William Sheehan, Associate Professor or Pediatrics, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAUSE-CNH-01; 1U01AI160090-01 (NIH)
Record Dates: First submitted 2022-03-30; First posted 2022-04-18 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Asthma in Children; Atopy; Viral Upper Respiratory Infection
MeSH Terms: conditions — Common Cold | interventions — Omalizumab

STUDY DESIGN:
Intervention Model Description: Single site, prospective, parallel-group, double-blinded, randomized clinical trial conducted over three consecutive fall seasons.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study site's research pharmacy will dispense the study drug as per the randomization schedule provided by REDCap. Prior to injection, an unblinded site pharmacist will confirm the expiration date, the dose, and randomization assignment. The injections will be administered in the Clinical Research Center at the study site by unblinded and trained nursing staff. The product will remain blinded to the investigators, other site staff, the participant, and legal guardians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omalizumab (Experimental): Single dose of omalizumab at the start of a viral upper respiratory infection as defined by onset of (or substantial worsening of) rhinorrhea, nasal congestion or sneezing (single or multiple symptoms) during the fall outcome season (defined as the 90-day period beginning on each child's return to school)
  Interventions: Drug: Omalizumab
- Placebo for omalizumab (Placebo Comparator): Single dose of placebo for omalizumab at the start of a viral upper respiratory infection as defined by onset of (or substantial worsening of) rhinorrhea, nasal congestion or sneezing (single or multiple symptoms) during the fall outcome season (defined as the 90-day period beginning on each child's return to school)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab — Omalizumab dose for each specific participant is based on that participant's weight and total IgE level. Omalizumab is provided by the manufacturer in two strengths:
  • For Injection: 75 mg/0.5 mL and 150 mg/mL solution in a single-dose prefilled syringe
  Other Names: Xolair
  Arms: Omalizumab
Drug: Placebo — Matching placebo for omalizumab will be provided in 0.5 mL and 1 mL solution for injection in pre-filled syringes.
  Other Names: Placebo for omalizumab
  Arms: Placebo for omalizumab

SUMMARY:
OBOE is a prospective, pilot, parallel group RCT with the overall aim of examining the effect of a single dose of anti-IgE (omalizumab) vs. placebo administered at the onset of URIs in the fall season among highly exacerbation-prone, urban, and atopic youth aged 6-17 years with persistent asthma. OBOE will recruit and randomize participants over 3 years (3 annual cohorts of participants). Recruitment for each of the yearly cohorts of OBOE will begin in February. Each cohort will be followed for a 2-6-month run-in period with the objective to gain control of each participant's asthma and to stabilize the required controller medication step level. Participants will receive routine asthma care every 1-2 months (a total of 2-4 times) during run-in using a previously described algorithm developed by the Inner-city Asthma Consortium and successfully employed in the PROSE study. The primary outcome is the change in the amount of nasal IFN-α recovered by nasal fluid absorption between two time points, within 72 hours of onset of a URI as defined by onset of (or substantial worsening of) rhinorrhea, nasal congestion or sneezing (single or multiple symptoms) and 3-6 days after study drug injection.

ELIGIBILITY:
Inclusion Criteria at Study Entry:

Participants must meet the following:

1. Parent or guardian must be able to understand and provide informed consent in English and participants ≥7 must be able to provide assent
2. 6-17 years, inclusive at time of screening
3. Physician-diagnosed persistent asthma
4. ≥1 exacerbation of asthma requiring systemic corticosteroids in the 6-month period before the planned start of the participant's upcoming school year or ≥2 exacerbations of asthma requiring systemic corticosteroids in the 12-month period before the planned start of the participant's upcoming school year
5. Sensitization to ≥1 perennial aeroallergen
6. Total serum IgE and weight appropriate for omalizumab dosing
7. Insurance that covers standard of care medications
8. Primary family residence (home where child sleeps a majority of nights) in a Metropolitan Statistical Area where ≥10% of families have income below poverty line and/or publicly funded health insurance
9. At least one of the following criteria:

   1. peripheral eosinophilia >300µL
   2. total serum IgE >300kU/L
   3. sensitization to ≥3 perennial aeroallergens
10. Females of childbearing potential must have a negative pregnancy test upon study entry
11. Females with reproductive potential must agree to use FDA approved methods of birth control for the duration of the study

Additional Inclusion Criteria (these must be met prior to randomization at the fall season sick visit A (SVa) during the 90-day outcome period):

In order to be eligible for randomization at the SVa visit, participants must also meet all of the following criteria:

1. Reporting onset of URI symptoms within 72 hours prior to SVa, confirmed by the study physician
2. Report no use of nasal corticosteroids or nasal vaccinations within 14 days prior to SVa
3. Have a negative rapid nasal swab antigen test for SARS-CoV-2
4. Be more than 14 days from the onset of any previous asthma exacerbation requiring systemic steroids
5. Have no current lower respiratory symptoms that, in the opinion of the study physician, require systemic corticosteroid treatment
6. Complete collection of nasal absorption sample within 72 hours of onset URI [defined by onset of (or substantial worsening of) rhinorrhea, nasal congestion or sneezing (single or multiple symptoms)] as determined by the study physician's assessment at the SVa visit

Exclusion Criteria:

1. Inability or unwillingness of a participant's parent or guardian to give written informed consent or comply with study protocol or inability or unwillingness of a participant ≥7 to provide assent
2. Contraindication to receipt of omalizumab
3. Presence of a second chronic medical condition (including but not limited to serious cardiorespiratory disorders, cancer, sickle cell disease, uncontrolled seizure disorder, auto-immune disorders, or type 1 diabetes)
4. Pregnancy or active lactation
5. History of latex allergy
6. Treatment with omalizumab or other monoclonal antibody, or aeroallergen immunotherapy in the prior six months
7. Plan for home schooling during the 90-day outcome period
8. History of life-threatening asthma defined by requirement for intubation or cardiorespiratory arrest
9. Inability of primary caregiver and child to speak English
10. In the opinion of the investigator, participant will not be able to wean from nasal steroids or to avoid nasal vaccinations during the 90-day fall outcome period
11. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Nasal interferon-α (IFN-α) | 3-6 day period after injection of study drug/placebo
  The change in the amount of nasal IFN-α recovered by nasal fluid absorption between two time points, when study drug/placebo is injected and 3-6 days later

SECONDARY OUTCOMES:
Nasal Type 2 Cytokines | 3-6 day period after injection of study drug/placebo
  Change in the amount of nasal type 2 cytokines recovered by nasal fluid absorption between two time points, when study drug/placebo is injected and 3-6 days later
Asthma Exacerbations | two weeks after injection of study drug/placebo
  Rate of exacerbations of asthma requiring systemic steroids in the two weeks following study drug/placebo injection.
Change in type 2 cytokine levels as a function of nasal airway microbiome | 3-6 day period after injection of study drug/placebo
  Change in type 2 cytokine levels between two time points (when study drug/placebo is injected and 3-6 days later) as a function of nasal airway microbiome phenotypes based on the abundance of Moraxella catarrhalis and Streptococcus pneumoniae and other microbial species recovered by nasal wash

OTHER OUTCOMES:
Local and systemic immune responses as measured by immune cellular phenotyping | 3-6 day period after injection of study drug/placebo
  To examine the effect of single-dose omalizumab vs placebo on nasal and systemic immune responses as measured by immune cellular phenotyping
Local and systemic immune responses as measured by gene expression profiling | 3-6 day period after injection of study drug/placebo
  To examine the effect of single-dose omalizumab vs placebo on nasal and systemic immune responses as measured by gene expression profiling
Local and systemic immune responses as measured by proteome | 3-6 day period after injection of study drug/placebo
  To examine the effect of single-dose omalizumab vs placebo on nasal and systemic immune responses as measured by proteome
Local and systemic immune responses as measured by metabolome | 3-6 day period after injection of study drug/placebo
  To examine the effect of single-dose omalizumab vs placebo on nasal and systemic immune responses as measured by metabolome
Asthma symptoms | 14 day period before sick visit C
  To examine the effect of single-dose omalizumab vs placebo on days of asthma symptoms in the prior 14 days
Albuterol use | 14 day period before sick visit C
  To examine the effect of single-dose omalizumab vs placebo on days of albuterol use in the prior 14 days
Asthma Control Test | 14-20 days after injection of study drug/placebo
  To examine the effect of single-dose omalizumab vs placebo on values derived from the Asthma Control Test
Pediatric Asthma Severity Score | 3-6 day period after injection of study drug/placebo
  To examine the effect of single-dose omalizumab vs placebo on the Pediatric Asthma Severity Score
Missed full school days | 14 day period before sick visit C
  To examine the effect of single-dose omalizumab vs placebo on missed full school days over the prior 14 days
Spirometry | 3-6 day period after injection of study drug/placebo
  To examine the effect of single-dose omalizumab vs placebo on spirometry parameters (FEV1, FVC, FEV1/FVC)
Unscheduled healthcare utilization (asthma-related urgent care visits, emergency department visits, hospitalizations) during the observation period | period from injection of study drug/placebo through study completion, a range of 60-150 days
  To examine the effect of single-dose omalizumab vs placebo on the rate of unscheduled healthcare utilization (asthma-related urgent care visits, emergency department visits, hospitalizations) during the post-randomization observation period (from injection to end of each participant's study participation)
Total Nasal Symptom Score | 14-20 days after injection of study drug/placebo
  To examine the effect of single-dose omalizumab vs placebo on the Total Nasal Symptom Score
Modified Rhinitis Symptoms Utility Index | 14 day period before sick visit C
  To examine the effect of single-dose omalizumab vs placebo on the Modified Rhinitis Symptoms Utility Index
Reliever medication usage (short acting beta agonists and systemic steroids) | period from injection of study drug/placebo through study completion, a range of 60-150 days
  To examine the effect of single-dose omalizumab vs placebo on reliever medication usage (short acting beta agonists and systemic steroids) during the post-randomization observation period (from injection to end of each participant's study participation)

CONTACTS AND LOCATIONS:
Overall Officials: William Sheehan, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No